CLINICAL TRIAL: NCT06588751
Title: Effects of SCALP Block on Postoperative Analgesia in Craniotomy Surgery: A Prospective, Randomized Controlled, Double-Blind Study
Brief Title: Effects of SCALP Block on Postoperative Analgesia in Craniotomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Muhammed Halit Satici, Specialist, Department of Anesthesiology, Konya City Hospital, M.D, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: scalp
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: After the surgical procedure, patients in Group S were placed in a semi-sitting position. Following skin antisepsis with 5% povidone-iodine, a sterile drape was applied. A circumferential scalp block with 2 cc of 0.25% bupivacaine was done on each of the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, greater occipital, and lesser occipital nerves that supply the forehead and scalp with sensory information. The procedure was performed bilaterally. The supratrochlear and supraorbital nerves were blocked at the brow, close to the upper middle edge orbit, and over the supraorbital notch that could be felt. The zygomaticotemporal nerve was blocked between the posterior edge of the zygomatic arch. The auriculotemporal nerve was blocked at the level of the tragus. The greater and lesser occipital nerves were blocked at the medial and lateral thirds of the superior nuchal line.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): After the surgery was completed, each patient received 3 mg of morphine IV and 8 mg of dexamethasone IV. Upon transfer to the intensive care unit, patients were administered 1 g of paracetamol IV three times a day and 20 mg of tenoxicam IV twice daily.
  Interventions: Other: Scalp block
- scalp block (Other): After the surgical procedure, patients in Group S were placed in a semi-sitting position. Following skin antisepsis with 5% povidone-iodine, a sterile drape was applied. A circumferential scalp block with 2 cc of 0.25% bupivacaine was done on each of the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, greater occipital, and lesser occipital nerves that supply the forehead and scalp with sensory information. The procedure was performed bilaterally. The supratrochlear and supraorbital nerves were blocked at the brow, close to the upper middle edge orbit, and over the supraorbital notch that could be felt. The zygomaticotemporal nerve was blocked between the posterior edge of the zygomatic arch. The auriculotemporal nerve was blocked at the level of the tragus. The greater and lesser occipital nerves were blocked at the medial and lateral thirds of the superior nuchal line.
  Interventions: Other: Scalp block

INTERVENTIONS:
Other: Scalp block — After the surgical procedure, patients in Group S were placed in a semi-sitting position. Following skin antisepsis with 5% povidone-iodine, a sterile drape was applied. A circumferential scalp block with 2 cc of 0.25% bupivacaine was done on each of the supraorbital, supratrochlear, zygomaticotemporal, auriculotemporal, greater occipital, and lesser occipital nerves that supply the forehead and scalp with sensory information. The procedure was performed bilaterally. The supratrochlear and supraorbital nerves were blocked at the brow, close to the upper middle edge orbit, and over the supraorbital notch that could be felt. The zygomaticotemporal nerve was blocked between the posterior edge of the zygomatic arch. The auriculotemporal nerve was blocked at the level of the tragus. The greater and lesser occipital nerves were blocked at the medial and lateral thirds of the superior nuchal line.

SUMMARY:
Patients undergoing craniotomy surgery often experience severe postoperative pain. This pain can affect the patient's hemodynamics, disrupt sleep patterns, and prolong hospital stays. Sudden increases in heart rate and blood pressure due to pain may lead to elevated intracranial pressure in patients, potentially causing morbidity and mortality. Opioids are commonly used to mitigate hemodynamic fluctuations and reduce postoperative pain; however, they may delay recovery, contribute to excessive sedation, and affect postoperative neurological examinations. Additionally, opioids have adverse effects such as nausea, vomiting, and respiratory depression. Alleviating hemodynamic instability and postoperative pain are critical concerns for neuro anesthesiologists. Regional analgesia techniques are employed in neurosurgery patients because they minimize anesthesia requirements, alleviate pain, and allow for neurological assessment with a lower incidence of systemic complications.The scalp block was developed due to its potential benefits as an effective regional anesthesia technique that supports the advancement of delicate brain surgeries such as functional and microsurgeries.

DETAILED DESCRIPTION:
In this study, we hypothesize that patients who receive a SCALP block will have lower postoperative Numerical Rating Scale scores and consume less total analgesia.

Our primary objective is to evaluate postoperative numerical rating scale scores in patients undergoing craniotomy surgery with a SCALP block.

Our secondary objectives are to assess the total amount of rescue analgesia consumed, the time to first rescue analgesia, patient satisfaction, and any possible complications. The study was planned as a prospective, randomized, controlled, double blind. At each clinic, an anesthesiologist randomly allocated patients to two significant groups using numbered opaque sealed envelopes: Group S (patients receiving SCALP block) and Group C (patients getting just multimodal analgesia). The anesthesiologists responsible for the randomization process were not involved in any other sections of the trial, and the individuals executing the SCALP blocks procedure were not engaged in other areas of the research. Additionally, the researcher who intervened, the participants, and the analyzer were blinded to the details of the study. After the surgery, two different anesthesia technicians recorded the primary and secondary results of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* General anesthesia
* American Society of Anesthesiologists physical status I-III

Exclusion Criteria:

* Contraindications to regional anesthesia
* Coagulation disorders
* Known allergy to local anesthetics
* Infections at the block site
* Pregnant patients
* Emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Scalp | One day
  Our primary objective is to evaluate postoperative numerical rating scale scores in patients undergoing craniotomy surgery with a SCALP block. (Numerical rating scale score 0-10 point. 0= Very Bad, 10= Very Good

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)